CLINICAL TRIAL: NCT07177612
Title: Implementation Research on the LILAC Method to Educate Management of Elevated Lipoprotein(a).
Acronym: LILAC-UNI
Status: Enrolling by invitation | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Loh Wann Jia, Primary Investigator (Senior consultant endocrinologist), Changi General Hospital
Other Study IDs: CIRB2025-0274
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lipoprotein(a); Lipoprotein(a), Hyper-Lp(a)-Emia
Keywords: LILAC-for-Lpa; Educational Videos; lipoprotein(a); Lp(a)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Professionals: This group includes participants who are doctors, nurses, pharmacists, allied health and healthcare related students
- Patients/Family/Public: This group includes participants who have high Lipoprotein(a) levels, or their family members, or members of the public.

SUMMARY:
The goal of this observational study is to assess the if short educational videos about #LILAC-for-Lpa are feasible and accepted in improving the confidence, testing, and management on Lipoprotein(a).

DETAILED DESCRIPTION:
The aims of this study are to (1) assess the feasibility of using these educational videos about LILAC-for-Lp(a) to help improve confidence, testing and the management of Lp(a), (2) assess the acceptability in using short education videos about LILAC-for-Lp(a) and (3) to understand the knowledge gaps of Lp(a) in medical professionals through the additional questionnaire provided.

ELIGIBILITY:
Inclusion Criteria:

* Participants include students, participants from institute of higher learning aged 16 and above.
* Participants aged 16 and above regardless of local or overseas, may also be from educational talks that Dr Loh is invited to speak at.
* Patients and members of the public aged 16 and above if they attend lipid awareness educational events.
* Participants aged 16 and above in patient support groups or patient advocacy networks.

Exclusion Criteria:

* Participants aged below 16 years old.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study populations include healthcare professionals, patients, and members of the public.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of Knowledge and awareness of Lp(a) | From enrolment to 3 months after
  Survey and questionnaire on participants to assess knowledge and awareness

SECONDARY OUTCOMES:
Acceptance of Educational Videos | From point of enrolment to 3 months
  Survey to determine if the educational videos are useful for them
Lipoprotein(a) Testing | During enrolment to 1 year
  Survey to doctors on whether they are testing for Lipoprotein(a) in their patients prior to watching the educational videos, 3 months after, and 1 year after.

CONTACTS AND LOCATIONS:
Locations (3):
- Online Portal, Australia, Perth, Australia
- Online web portal, Kuala Lumpur, Malaysia
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
This is an educational research survey

REFERENCES:
- [Background] Loh WJ, Pang J, Simon O, Chan DC, Watts GF. Deficient perceptions and practices concerning elevated lipoprotein(a) among specialists in Singapore. Front Cardiovasc Med. 2025 Feb 14;12:1527351. doi: 10.3389/fcvm.2025.1527351. eCollection 2025. PMID 40027516
- [Background] Loh WJ, Watts GF, Lum E. A short educational video for improving awareness and confidence of healthcare professionals in managing lipoprotein(a): a pilot study based on LILAC-for-Lp(a). Eur J Cardiovasc Nurs. 2025 Jul 21;24(5):796-799. doi: 10.1093/eurjcn/zvaf052. No abstract available. PMID 40156158